CLINICAL TRIAL: NCT02179190
Title: Prospective, Multi-Center, Single-Arm Study of Reverse Medical Barrel™ Vascular Reconstruction Device for Adjunctive Treatment to Embolic Coils in Wide-Neck, Intracranial, Bifurcating Aneurysms of Middle Cerebral and Basilar Arteries
Brief Title: Reverse Medical Barrel™ Device for Adjunctive Treatment for Wide-Neck, Intracranial, Bifurcating/Branching Aneurysms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Neurovascular Clinical Affairs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VRD-001
Record Dates: First submitted 2014-06-27; First posted 2014-07-01 (Estimated); Results first posted 2018-12-05 (Actual); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Intracranial Bifurcating Aneurysms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- BARREL VRD (Experimental): The Barrel VRD was implanted as adjunctive to embolic coils in subjects with wide necked bifurcating aneurysms within the Middle Cerebral and Basilar Arteries.
  Interventions: Device: BARREL VRD

INTERVENTIONS:
Device: BARREL VRD — The Barrel VRD was implanted as adjunctive to embolic coils in subjects with wide necked bifurcating aneurysms within the Middle Cerebral and Basilar Arteries.

SUMMARY:
Single arm study to evaluate the outcomes of treatment with the Barrel VRD device as an adjunctive treatment to coiling for wide neck, intracranial, bifurcating/branching aneurysms in the middle cerebral and basilar arteries.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between 18 and 85 years old.
2. A wide-neck de novo or non-de novo aneurysm.
3. Appropriate informed consent obtainable as determined by local IRB.
4. Life expectancy > 24 months.

Exclusion Criteria:

1. Aneurysm rupture within 30 days of enrollment.
2. Bifurcating aneurysms not treatable with coiling.
3. Subject has platelet count of <70,000.
4. Subject has known allergies to nickel-titanium metal.
5. Subject has known allergies to aspirin or heparin.
6. Subject has a life-threatening allergy to contrast (unless treatment for allergy can be tolerated).
7. Subject is currently participating in another clinical research study.
8. Subject is pregnant or breastfeeding.
9. Subject has participated in a drug study within the last 30 days.
10. Subject is unable or unwilling to comply with protocol requirements and obtain required clinical evaluations and follow-up.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2014-10-13 (Actual); Primary Completion 2017-07-21 (Actual); Study Completion 2017-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J Mocco, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (3):
- United States (3):
  - Baptist Medical Center Jacksonville, Jacksonville, Florida
  - Baptist Hospital of Miami, BCVI, Miami, Florida
  - Tallahassee Neurological Clinic, Tallahassee, Florida

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- BARREL VRD: The Barrel VRD was implanted as an adjunctive to embolic coils in subjects with wide necked bifurcating aneurysms within the Middle Cerebral and Basilar Arteries. BARREL VRD: The Barrel VRD was implanted as adjunctive to embolic coils in subjects with wide necked bifurcating aneurysms within the Middle Cerebral and Basilar Arteries.
Period: Enrollment
Arm/Group | BARREL VRD
Started (Participants Consented and Assessed for Eligibility) | 138
Completed (Attempted with the Study Device - Intent to Treat Population) | 127
Not Completed | 11
Not completed — Exit Prior to Device Attempt | 11
Period: Index Procedure With Barrel VRD Attempt
Arm/Group | BARREL VRD
Started (Participants with an attempted Barrel VRD Implant) | 127
Completed (Participants with a Successful Barrel Implant) | 120
Not Completed | 7
Not completed — Did not receive Barrel VRD | 7
Period: Follow-Up Post Barrel VRD Implanted
Arm/Group | BARREL VRD
Started (Participants Implanted with the Barrel VRD Expected to Complete the 12 Month Visit) | 120
Completed (Participants Implanted with the Barrel VRD that Completed the 12 Month Visit) | 111
Not Completed | 9
Not completed — Death | 3
Not completed — Withdrawal by Subject | 3
Not completed — Physician Decision | 2
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Participants with enrolled (consented ) with an attempted Barrel VRD Implant
Arm/Group | BARREL VRD
Number analyzed (Participants) | 127
Age, Continuous [Mean (Standard Deviation); unit: years]
  Mean ± Standard Deviation | 60.4 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91
  Male | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12
  Not Hispanic or Latino | 108
  Unknown or Not Reported | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 108
  More than one race | NA — Subjects with more than one race were not collected
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Neurologic Death or Major Ipsilateral Stroke Within 12 Month Follow-up Period.
Description: The primary safety endpoint was the number of participants reported with a neurological death or major ipsilateral stroke (National Institute of Stroke Scale (NIHSS) increase of ≥ 4 for > 24 hours) at any time during the follow-up period.
  The NIHSS is a tool used to quantify neurological impairment caused by stroke. The scale interpretation is as follows:
  0: No stroke symptoms 1-4: Minor stroke symptoms 5-15: Moderate stroke 16-20: Moderate to severe stroke 21-42: Severe strokeThe National Institutes of Health Stroke Scale
Time Frame: 12 months, after device implant
Population: Participants implanted with the Barrel VRD
Measure: Count of Participants; unit: Participants
Arm/Group | BARREL VRD
Number analyzed (Participants) | 127
Participants | 5

2. Primary Outcome: Number of Participants With Raymond Grade I ( 100%) Occlusion of the Aneurysms for Participants Treated With the Barrel VRD at 12 Months in the Absence of Retreatment, Parent Artery Stenosis, or Target Aneurysm Rupture
Description: The primary effectiveness endpoint was the count of participants achieving Raymond Grade I (100% occlusion) of the aneurysm treated with the Barrel VRD at 12 months ± 8 weeks in the absence of retreatment, parent artery stenosis (>50%), or target aneurysm rupture
  The Raymond Grade Classification definitions evaluated by an independent core laboratory are as follows:
  Class 1: Complete occlusion - complete obliteration of the aneurysm. Class 2: Residual neck - persistence of any portion of the original defect of the arterial wall as seen on any single projection, but without opacification of the aneurysmal sac.
  Class 3: Residual aneurysm - opacification of the aneurysmal sac
Time Frame: 12 months, after device implant
Population: Subjects treated with the Barrel VRD that completed the 12 month visit imaging
Measure: Count of Participants; unit: Participants
Arm/Group | BARREL VRD
Number analyzed (Participants) | 106
Participants | 67

3. Secondary Outcome: Number of Participants With Successfully Deployed Barrel VRD
Description: This secondary outcome measure provides the number of subjects successfully implanted with the Barrel VRD.
Time Frame: Index Procedure, Day 0
Measure: Count of Participants; unit: Participants
Arm/Group | BARREL VRD
Number analyzed (Participants) | 127
Participants | 120

4. Secondary Outcome: Number of Participants With Raymond Grade I (100% Complete Occlusion) and Raymond Grade II (Residual Neck) for Participants Treated With the Barrel VRD, in the Absence of Retreatment, Parent Artery Stenosis (>50%), or Target Aneurysm Rupture at 12 Months
Description: This secondary outcome measure provides the count of participants treated with the Barrel VRD with Independent Core Laboratory aneurysm occlusion imaging evaluations of Complete Occlusion (Raymond Grade I) and Residual Aneurysm Neck (Raymond Grade II) at 12 months combined. Subjects with evidence of parent artery stenosis, retreatment, or rupture were not considered success.
  Raymond Grade Scale
  Class 1: Complete occlusion - complete obliteration of the aneurysm. Class 2: Residual neck - persistence of any portion of the original defect of the arterial wall as seen on any single projection, but without opacification of the aneurysmal sac.
  Class 3: Residual aneurysm - opacification of the aneurysmal sac.
Time Frame: 12 months, after device implant
Population: Outcomes are based on observed data (i.e., 106 participants with 12-month evaluable imaging). 21/127 participants did not have evaluable imaging at 1-Year.
Measure: Count of Participants; unit: Participants
Arm/Group | BARREL VRD
Number analyzed (Participants) | 106
Participants | 75

5. Secondary Outcome: Number of Participants With Modified Rankin Score of 0-2 or no Change From Baseline
Description: This secondary outcome provides the count of participants treated with the Barrel device with a Modified Rankin Score of 0-2 at 12 months or no change from baseline.
  The Modified Rankin Score is a scale for measuring general functionality as follows:
  0: No symptoms at all
  1. No significant disability despite symptoms; able to carry out all usual duties and activities
  2. Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance
  3. Moderate disability; requiring some help, but able to walk without assistance
  4. Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance
  5. Severe disability; bedridden, incontinent and requiring constant nursing care and attention
  6. Dead
Time Frame: 12 months, after device implant
Population: Outcomes are based on observed data, from 111 participants completed at 1-year and 3 participants with an mRS score of 6 (death) prior to 1 year.
Measure: Count of Participants; unit: Participants
Arm/Group | BARREL VRD
Number analyzed (Participants) | 114
Participants | 107

6. Secondary Outcome: Number of Participants With Angiographic Evidence of In-stent Stenosis at 12 Months +/- 8 Weeks Reported According to the Following Ordinal Groups: <25%, 25-50%, 51-75%, >75%
Description: This secondary measure provides the count of participants with parent artery stenosis per an independent core lab evaluation within the following ordinal groups: <25%, 25-50%, 51-75%, >75%.
Time Frame: At 12 Months +/- 8 weeks
Population: Outcomes are based on observed data on 89 participants with evaluable angiographic data at 1 year. 38/127 participants did not have angiographic data at 1 year available for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | BARREL VRD
Number analyzed (Participants) | 89
Participants
  In-Stent Stenosis at 12 Months < 25% | 88
  In-Stent Stenosis at 12 Months 25-50% | 1
  In-Stent Stenosis at 12 Months 51-75% | 0
  In-Stent Stenosis at 12 Months < 75% | 0

7. Secondary Outcome: Number of Participants With Any Cause of Death Within 30 Days or Neurological Death Within 12 Months +/- 8 Weeks
Description: This secondary outcome measure provides the combined number and percentage of subjects that died within 30 days or had a neurologic death within 12 months of receiving the study device.
Time Frame: 30 Days and 12 months +/- 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | BARREL VRD
Number analyzed (Participants) | 127
Participants | 1

8. Other Pre Specified Outcome: Number of Participants With Reported Device Related Serious Adverse Events
Description: This secondary outcome measure provides the count of participants reported with a Serious Device Related Adverse Events
Time Frame: From the point of consent until participant exits the study at 1 year
Population: Subjects with an Attempted Barrel VRD Implant
Measure: Count of Participants; unit: Participants
Arm/Group | BARREL VRD
Number analyzed (Participants) | 127
Participants | 4

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from the point of consent through the study exit at 12 months.
Description: The adverse event data reported by sites was adjudicated by a three member independent Clinical Events Committee (CEC). All data presented within this section has been CEC adjudicated. Adjudicable events met the following criteria:
  * Neurological cause adverse events with a corresponding worsening of NIHSS,
  * All Device related adverse events,
  * All Procedure related adverse events,
  * All SAEs, and
  * All Antiplatelet therapy related events.
Arm/Group | BARREL VRD
All-Cause Mortality (participants affected / at risk) | 3/127
Serious Adverse Events (participants affected / at risk) | 44/127
Other Adverse Events (participants affected / at risk) | 73/127
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BARREL VRD (N=127)
Anaemia (Blood and lymphatic system disorders) | 4 (4)
Acute myocardial infarction (Cardiac disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 2 (2)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (1)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 2 (2)
Adverse drug reaction (General disorders) | 1 (1)
Catheter site haematoma (General disorders) | 2 (2)
Pneumonia bacterial (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 3 (3)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Retroperitoneal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Brain oedema (Nervous system disorders) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 1 (1)
Cerebral infarction (Nervous system disorders) | 2 (2)
Convulsion (Nervous system disorders) | 2 (2)
Haemorrhage intracranial (Nervous system disorders) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (2)
Hydrocephalus (Nervous system disorders) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 8 (8)
Migraine (Nervous system disorders) | 1 (1)
Status epilepticus (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Vertebral artery dissection (Nervous system disorders) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1)
Glomerulonephritis rapidly progressive (Renal and urinary disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Spinal decompression (Surgical and medical procedures) | 1 (1)
Aneurysm (Vascular disorders) | 1 (1)
Hypertensive emergency (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BARREL VRD (N=127)
Catheter site haemorrhage (General disorders) | 7 (7)
Headache (Nervous system disorders) | 24 (27)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Ecchymosis (Skin and subcutaneous tissue disorders) | 9 (10)
Palpitations (Cardiac disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Diplopia (Eye disorders) | 1 (1)
Eyelid ptosis (Eye disorders) | 2 (2)
Photopsia (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 3 (4)
Visual impairment (Eye disorders) | 3 (3)
Colitis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 9 (9)
Oral mucosal blistering (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Catheter site haematoma (General disorders) | 5 (5)
Catheter site inflammation (General disorders) | 1 (1)
Catheter site swelling (General disorders) | 1 (1)
Chest pain (General disorders) | 2 (2)
Drug intolerance (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Injection site haemorrhage (General disorders) | 1 (1)
Local swelling (General disorders) | 1 (1)
Thrombosis in device (General disorders) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1)
Procedural hypertension (Injury, poisoning and procedural complications) | 1 (1)
Procedural hypotension (Injury, poisoning and procedural complications) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1)
Radiation skin injury (Injury, poisoning and procedural complications) | 1 (1)
Wound secretion (Injury, poisoning and procedural complications) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 1 (1)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Amnesia (Nervous system disorders) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1)
Balance disorder (Nervous system disorders) | 1 (1)
Cerebral artery thrombosis (Nervous system disorders) | 2 (2)
Cerebral infarction (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 7 (8)
Hypoaesthesia (Nervous system disorders) | 2 (3)
Migraine (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 2 (2)
Spondylitic myelopathy (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 3 (4)
Tremor (Nervous system disorders) | 1 (1)
Disorientation (Psychiatric disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Urethral pain (Renal and urinary disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Aneurysm repair (Surgical and medical procedures) | 1 (1)
Aneurysm (Vascular disorders) | 1 (1)
Arterial stenosis (Vascular disorders) | 3 (3)
Intermittent claudication (Vascular disorders) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1)
Vasospasm (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-18): https://cdn.clinicaltrials.gov/large-docs/90/NCT02179190/Prot_SAP_000.pdf